CLINICAL TRIAL: NCT00369746
Title: Treatment of Depression Concurrent With Alcohol Abuse, an Extension of Alcohol Use Disorder in Patients Treated for Depression
Brief Title: STAR*D Alcohol: Treatment of Depression Concurrent With Alcohol Abuse
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: #5173; R01AA013303 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2011-12

CONDITIONS: Major Depressive Disorder; Alcohol Use Disorder
Keywords: Depression; Alcohol Abuse; Alcohol Dependence
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism; Depression | interventions — Citalopram

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alcohol and major depression, citalopram: Patients with alcohol use disorder and major depression, treated with citalopram tablets, 20-60 mg, once daily, for 12 weeks
  Interventions: Drug: citalopram
- Major Depression, citalopram: Patients with major depression, treated with citalopram tablets 20-60 mg daily, for 12 weeks
  Interventions: Drug: citalopram

INTERVENTIONS:
Drug: citalopram — tablets, 60 mg maximum, daily, 12 weeks
  Other Names: Celexa

SUMMARY:
The purpose of this study is to determine if having an alcohol use disorder affects recovery from depression, and also whether recovery from depression in patients who have alcohol use disorders is also accompanied by improvement in the alcohol use disorder.

DETAILED DESCRIPTION:
This is an extension of the multi-site sub-study of the National Institute of Mental Health (NIMH) protocol, Sequenced Treatment Alternatives to Relieve Depression (STAR*D), which utilized the infrastructure of the Depression Trials Network to enroll 4,000 subjects diagnosed with Major Depressive Disorder. These subjects initially received 12 weeks of treatment with the anti-depressant citalopram. The thrust of this study was to test treatment algorithms for those subjects who did not respond adequately to initial monotherapy treatment with citalopram or who were unable to tolerate it. The parent protocol also contained several ancillary studies, including a sub-study of subjects with co-morbid alcohol use disorders, which enrolled 130 subjects. Treatment response data was collected at multiple intervals during the 12 week treatment period on depressed subjects both with and without a co-morbid alcohol use disorder.

Comparison: Treatment outcome measures of subjects diagnosed with Major Depressive Disorder will be compared to treatment outcome measures of subjects diagnosed with Major Depressive Disorder and an Alcohol Use Disorder following the initial 12 week citalopram treatment period. This comparison will show whether having a co-morbid alcohol use disorder affects recovery from depression. In addition, alcohol use data of depressed subjects who demonstrated a positive response to anti-depressant treatment will be compared with alcohol use data of depressed subjects who did not have positive treatment outcomes. This comparison will show whether recovery from depression is associated with improvement in the co-morbid alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18- 75 years
* Meets criteria for Non-psychotic Major Depression
* Signs informed consent and able to comply with study
* Hamilton Depression Scale (HAM-D 17) >14
* Endorses any drinking items on Short Michigan Alcoholism Screening Test

Exclusion Criteria:

* Pregnant women and women of childbearing potential who are not using a medically accepted means of contraception.
* Women who are breast feeding
* Patients with suicidal ideation that require hospitalization
* Patients with unstable physical disorders
* Patients with a history of allergy to citalopram or history of non-response to an adequate dose of citalopram in the current episode.
* Patients meeting criteria for the following diagnoses as a primary condition: Schizophrenia, Schizoaffective Disorder, Bipolar I, II, and Not Otherwise Specified, Anorexia nervosa, Bulimia, Obsessive Compulsive Disorder
* Patients abusing substances which require detoxification. American Society for Addiction Medicine standards for detoxification will be used (Level III.7). Patients with substance abuse who are in substance abuse treatment will be eligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the Sequenced Treatment Alternatives to Relieve Depression
Sampling Method: Non-Probability Sample
Enrollment: 674 (Actual)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. McGrath, MD, Study Director — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from all participants entering the Sequenced Treatment Alternatives to Relieve Depression clinical trial.
Groups:
- Alcohol Abuse or Dependence: Subjects with alcohol abuse or dependence and Major Depression
- Major Depression Only: Major Depression without alcohol abuse disorder
Period: Overall Study
Arm/Group | Alcohol Abuse or Dependence | Major Depression Only
Started | 138 | 536
Completed | 138 | 536
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alcohol Abuse or Dependence: Subjects with alcohol abuse or dependence
- Total: Total of all reporting groups
Arm/Group | Alcohol Abuse or Dependence | Major Depression Only | Total
Number analyzed (Participants) | 138 | 536 | 674
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 138 | 536 | 674
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (12.3) | 39.5 (13.4) | 38.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 134 | 211
  Male | 61 | 402 | 463
Region of Enrollment [Number; unit: participants]
  United States | 138 | 536 | 674

OUTCOME MEASURES:

1. Primary Outcome: Quick Inventory of Depression- Self Report 16
Description: Quick Inventory of Depression- Self Report assesses 16 depressive symptoms experienced in the past week, based on self-rating, measured at study exit visit
  Scale range:
  Each of the four possible answers to each quiz is given an ascending numerical value from 0 to 3, and the total test score is the sum of the following: The highest number from questions 1-4 The number from question 5 The highest number from questions 6-9 The total of each question from 10-14 The highest number from questions 15-16
  Total scoring ranges (0-48):
  0-5, No Depression Likely 6-10, Possibly Mildly Depressed 11-15, Moderate Depression 16-20, Severe Depression 21 or Over, Very Severe Depression
Time Frame: study exit visit, at Week 12
Population: All participants who met entry criteria for alcohol abuse or dependence per protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Alcoholic: Subjects with alcohol abuse or dependence
- Major Depression Only: citalopram (Non alcoholic)
Arm/Group | Alcoholic | Major Depression Only
Number analyzed (Participants) | 138 | 536
units on a scale | 9.3 (6.1) | 8.9 (5.7)

2. Secondary Outcome: Timeline Follow Back (TLFB) Average Drinks Per Drinking Day
Description: This variable reports average drinks/drinking day in a pre-defined time frame.
Time Frame: 30 days
Population: Subjects who met entering criteria for alcohol abuse or alcohol dependence per protocol
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | Alcoholic
Number analyzed (Participants) | 138
drinks per drinking day | 2.9 (2.6)

3. Secondary Outcome: Quantitative Substance Use Inventory ((SUI)
Description: Quantitative Substance Use Inventory ((SUI) Measure substance use
  Administered at either week 12 or 14: Any Illicit Drug Using in last 30 days
Time Frame: 30 days
Population: All participants who met entry criteria for alcohol abuse or dependence per protocol.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Alcoholic
Number analyzed (Participants) | 138
Days | 2.4 (7.12)

4. Secondary Outcome: Timeline Follow Back (TLFB) Drinking Days Per 30 Days
Description: This variable reports drinking days in a pre-defined time frame.
Time Frame: 30 days
Population: Subjects who met entering criteria for alcohol abuse or alcohol dependence per protocol
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Alcoholic
Number analyzed (Participants) | 138
days | 8.1 (7.8)

5. Secondary Outcome: Timeline Follow Back (TLFB) Maximum Drinks Per Drinking Day
Description: This variable reports maximum drinks per drinking day in a pre-defined time frame.
Time Frame: 30 days
Population: Subjects who met entering criteria for alcohol abuse or alcohol dependence per protocol
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | Alcoholic
Number analyzed (Participants) | 138
drinks | 4.9 (3.9)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Alcohol Abuse or Dependence | Major Depression Only
Serious Adverse Events (participants affected / at risk) | 8/138 | 23/536
Other Adverse Events (participants affected / at risk) | 0/138 | 0/536
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alcohol Abuse or Dependence (N=138) | Major Depression Only (N=536)
Hospitalilization GMC (General disorders) | 5 (5) | 16 (16)
Medical illness without hospitalizaiton (General disorders) | 1 (1) | 1 (1)
Psychiatric hospitalization, substance abuse (Psychiatric disorders) | 2 (2) | 1 (1)
Death, non-suicide (General disorders) | 0 (0) | 1 (1)
Psychiatric hospitalization (worsening depression) (Psychiatric disorders) | 0 (0) | 2 (2)
Psychiatric hospitalization (Other) (Psychiatric disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes